CLINICAL TRIAL: NCT07075692
Title: Effects of Physiotherapy Applications in Children With Bladder and Bowel Symptoms After Anorectal Malformation Surgery
Brief Title: Physiotherapy Applications in Children With Bladder and Bowel Symptoms After Anorectal Malformation Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, Professor, Ankara Yildirim Beyazıt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1328
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Anorectal Diseases
MeSH Terms: conditions — Rectal Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy group (Experimental): Physiotherapy program will be performed
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy program will include patient education, lifestyle recommendations (fluid intake, diet, correct urination/defecation position, weight control, etc.), breathing exercises, pelvic floor muscle training, and stabilization exercises. The treatment program will last for a total of 8 weeks

SUMMARY:
The aim of our study was to investigate the effects of physiotherapy applications in children with bladder and bowel symptoms after anorectal malformation surgery.

DETAILED DESCRIPTION:
Anorectal malformation (ARM) is a congenital anomaly in which the rectum and anus of the developing fetus fail to form normally before birth. The main treatment for ARM is surgery. However, various complications may occur in these children after surgery due to disruption of the muscular structure, nerve damage and weakness of the sphincters. These complications include fecal incontinence, chronic constipation, difficulty in defecation and abdominal pain. Constipation and fecal incontinence can be seen quite frequently in these individuals. Sometimes these symptoms may be accompanied by additional bladder problems (urinary incontinence etc.). Bowel training, dietary recommendations, toilet training, enemas, medications and physiotherapy applications can be used in the management of fecal incontinence and constipation. In the literature, there are limited number of studies evaluating physiotherapy applications in the management of postoperative bladder bowel symptoms in children with ARM.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 years with bladder bowel symptoms after anorectal malformation surgery
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of a congenital and/or chronic disease
* Having a history of any additional neurological, orthopedic or psychiatric disease that will affect the evaluation parameters
* Mental retardation
* Having received physiotherapy within the last 1 year

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Bladder and Bowel Dysfunction Symptoms | before and after treatment (8-week change)
  Bladder and bowel symptoms will be assessed with the Bladder and Bowel Dysfunction Score. The scale consists of 14 questions. The total score ranges from 0-52 and an increase in score means an increase in symptom severity.

SECONDARY OUTCOMES:
Bowel Function | before and after treatment (8-week change)
  Bowel function will be evaluated with a bowel diary. They will be asked to keep a bowel diary for 1 week, including the number and type of daily stools and the number of incontinent stools.
Bladder function | before and after treatment (8-week change)
  Bladder function will be evaluated with bladder diaries including voiding frequency, voiding volüme and number of incontinence In the bladder diary, they will be asked to fill in a 3-day bladder diary.
Constipation | before and after treatment (8-week change)
  Children's constipation will be evaluated with the Rome IV criteria. These criteria include; two or less defecation per week, fecal incontinence at least once a week, history of holding/ delaying the large toilet, painful and difficult bowel movements, presence of large feces in the rectum, presence of a history of large feces that can block the toilet
Pelvic floor muscle function | before and after treatment (8-week change)
  Pelvic floor muscle function will be evaluated with palpation form anus. The presence of correct contraction and relaxation of the pelvic floor muscle will be determined.
Life quality | before and after treatment (8-week change)
  Quality of life will be assessed with the Pediatric Quality of Life Inventory (PedsQL). The PedsQL consists of 23 items. It are scored between 0-100. The higher the total score of the quality of life, the better health-related quality of life is perceived.
Perception of improvement | after treatment (8-week change)
  Subjective perception of improvement will be assessed as -1 (worse), 0 (no change) and 1 (better).
Compliance with recommendations | After treatment (8-week change)
  Compliance with post-treatment recommendations will be assessed with the Visual Analog Scale (VAS). The VAS is a horizontal line with "0" at one end as "never compliance" and '10' at the other end as "always compliance".